CLINICAL TRIAL: NCT00448955
Title: A Phase III Open-Label Study of the Efficacy and Safety of ARD-0403, a Testosterone Cream, in Testosterone Deficient Men
Brief Title: Open-Label Study of ARD-0403 in Testosterone Deficient Men
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ardana Bioscience Ltd (Industry)
Responsible Party: Ardana Bioscience Ltd., Ardana Bioscience Ltd.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARD-0403-004
Record Dates: First submitted 2007-03-16; First posted 2007-03-19 (Estimated); Last update posted 2008-04-18 (Estimated); Status verified 2008-04

CONDITIONS: Hypogonadism
MeSH Terms: conditions — Hypogonadism

INTERVENTIONS:
Drug: ARD-0403 — ARD-0403

SUMMARY:
Male hypogonadism, a disorder associated with testosterone deficiency, is frequently seen in clinical practice and has significant effects on patient wellbeing. The purpose of this study is to investigate the efficacy and safety of ARD-0403 as a testosterone replacement therapy in testosterone deficient men.

ELIGIBILITY:
Inclusion Criteria:

* Testosterone deficiency

Exclusion Criteria:

* Previous treatment with testosterone replacement therapy within 4 weeks
* Moderate-severe benign prostatic hypertrophy, or prostatic cancer
* Haematocrit >50%

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic

SECONDARY OUTCOMES:
Safety and tolerability

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Medical Affiliated Research Center, Inc, Huntsville, Alabama
  - Stanford University, Stanford, California
  - Los Angeles Biomedical Research Institute at Harbor-UCLA, Torrance, California
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Michael E. Debakey VAMC, Houston, Texas
  - dgd Research, San Antonio, Texas
  - VA Puget Sound Health Care System, Seattle, Washington